CLINICAL TRIAL: NCT06468189
Title: Clinical and Neurophysiological Effects of Simultaneous Application of tDCS to Visual and Motor Cortex in Migraine; Double Blind Randomized Controlled Study
Brief Title: Clinical and Neurophysiological Effects of tDCS to Visual and Motor Cortex in Migraine
Acronym: MIRAGE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Alanya Alaaddin Keykubat University (Other); Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Prof. Lutfu Hanoglu, MD, Prof. Dr., Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023IMU_Migraine_tDCS
Record Dates: First submitted 2024-03-04; First posted 2024-06-21 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2024-06

CONDITIONS: Migraine
Keywords: transcranial direct current stimulation; tDCS; migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tDCS (Experimental): tDCS Interictal application will be performed during the attack-free period. Experimental group, 3 consecutive sessions, cathodal to occipital cortex (O1 or O2, ipsilateral); anodal to M1 (left)
  Interventions: Device: transcranial direct stimulation
- Sham (Sham Comparator): Control group, 3 consecutive sessions of sham stimulation to the same locations.
  Interventions: Device: Sham treatment

INTERVENTIONS:
Device: transcranial direct stimulation — Mars-01(Marslab, Turkey) transcranial direct current stimulation device works with a 9 volt battery and consists of two 5x5 (25 cm2) electrodes (anode and cathode). 3 consecutive sessions (days), cathodal to occipital cortex (O1 or O2, ipsilateral); Anodal application will be made to M1 (left). Active stimulation is 2mA tDCS with a 0 to 30 second acceleration period of 20 minutes per session. Placebo stimulation will be applied according to the device's own sham software protocol. Accordingly, the current consists of 30 seconds of increase from 0 to 2mA(milliamp), 10 seconds of stimulation, 30 seconds of decrease to 0 and 20 minutes of current-free application.
  Arms: tDCS
Device: Sham treatment — The same device used for stimulation will be used, but no stimulation will be given.
  Arms: Sham

SUMMARY:
tDCS can be offered as an alternative to migraine patients who have frequent and severe attacks and who are resistant to or unresponsive to preventive drug therapy. Additionally, this technique may also be an option for patients who refuse or have contraindications to taking anti-migraine medications. A decrease in headache severity and frequency is expected with this neuromodulation applied to migraine patients with frequent attacks. Based on this hypothesis; This tested whether simultaneous modulation of motor (M1, left) and visual cortex (O1 or O2, ipsilateral) with tDCS applied for 3 consecutive days is an effective treatment for migraine patients for the following specific purposes . No significant undesirable effects are expected, except for possible side effects that are simple and do not require medical intervention, such as tingling or itching in the area where the electrodes are attached, moderate fatigue, mild headache, nausea at a rate of less than 3%, and insomnia at a rate of less than 1%. . The research will be conducted within the framework of ethical principles and in accordance with the good clinical practice protocol.

A) The primary purpose of this study is to determine whether transcranial direct current stimulation applied simultaneously to the motor and visual cortex in migraine patients provides a significant reduction in pain due to migraine attacks compared to sham tDCS. Additionally, to evaluate the effects of this treatment, They will be measured changes in the number of migraine attacks, abortive medication intake (e.g., opioids, triptans), as well as overall improvement in cognitive status and quality of life. In addition, electrophysiological EEG evaluations, before and after treatment, and the results of these measurements, as a potential biomarker in migraine, will be compared in the active and sham groups.

B) It is aimed to determine whether the clinical effects of tDCS are long-lasting. Therefore, It will compared whether there is a difference in improvement of migraine-related pain between active and sham tDCS at pre-treatment (baseline) assessments as well as at 1, 2, and 3 months after treatment.

C) Finally, it will be examined whether tDCS treatment applied for 3 consecutive days in migraine patients is safe. Safety will be evaluated through neuropsychological testing and adverse event reporting.

DETAILED DESCRIPTION:
Headache disorders are quite common. In the 2016 Global Burden of Disease Study, migraine was the second highest cause of disability overall and the most common disease causing disability in young adults (15-49 years). When there are frequent or severe migraine attacks, pharmacological agents are used to reduce the frequency of migraine attacks. Standard migraine prophylactic treatments show either low efficacy or undesirable side effects, and most of them are licensed for other diseases and not for migraine. Additionally, some migraine patients are hesitant to choose pharmacological treatment. Compliance with these treatments is also quite low in the medication-using group. Recently used calcitonin gene-related peptide (CGRP) monoclonal antibody treatments are quite expensive treatments. Therefore, there remains a need for an effective, tolerable and affordable prophylactic treatment for migraine.

Migraine is complex, involving several circuits of both the central and peripheral nervous system and has a still unclear pathophysiology. Trigeminovascular activation is the key event of migraine pain, mostly related to the peripheral nervous system, but the central nervous system also plays a role in the formation and perception of migraine. The cerebral cortex of migraineurs is hypersensitive (overexcitable) to external stimuli, possibly due to altered functional connectivity in subcortical structures, including the thalamus. This resulting "thalamo-cortical dysrhythmia" and changes in excitability can be controlled with non-invasive neuromodulation techniques such as transcranial magnetic stimulation (TMS) and transcranial direct current stimulation (tDCS).

Non-invasive neuromodulation is applied to various forms of primary headaches and is recommended as an easily applicable method for both episodic and chronic migraine. So far, only single pulse transcranial magnetic stimulation (sTMS), vagus nerve stimulation (VNS), and supraorbital neurostimulation have been approved by the FDA for the treatment of migraine. Transcranial direct current stimulation (tDCS; direct current stimulation) is an electrical stimulation method used for non-invasive brain stimulation, where a weak electrical current of approximately 2 milliamps is applied through two scalp electrodes with a portable battery-powered system. tDCS is an electrical stimulation technique in which low-amplitude direct current is applied to the skull via surface electrodes, thereby modulating neural brain activity. The applied current changes the transmembrane neuronal potential and thus affects the level of excitability. Depending on the polarity of the active electrodes, tDCS can increase or decrease cortical excitability. tDCS has been shown to trigger changes in neuropsychological and motor activity in the brain. Protocols with variable session numbers (1-20 days) applied to different targeted brain regions provide promising results in pain syndromes by regulating pain-related pathways in various ways. Stimulation of the motor cortex with tDCS has already been shown to relieve pain in patients with traumatic spinal cord injury and other chronic pain syndromes, including fibromyalgia. Migraine patients are often hypersensitive to pain. A treatment that targets areas of the brain involved in the experience of pain may also help reduce pain in migraine patients. According to the results of systematic review and meta-analysis of studies conducted so far; tDCS has been evaluated as an effective, reliable method that can improve migraine symptoms by activating the motor cortex or activating/inhibiting the visual cortex. Additionally, tDCS treatment repeated for days over a period of 4 weeks or longer is effective in reducing migraine pain severity and attack duration. The benefit of tDCS may persist for at least 4 weeks after completion of the last tDCS session. Both anodal and cathodal stimulation have been evaluated as effective for reducing migraine pain severity. The study protocol present here aims to test a unique protocol with simultaneous anodal stimulation to the motor area and cathodal stimulation to the visual cortex. In the meta-analyses conducted so far; In future clinical studies using tDCS in migraine, the importance of simultaneously measuring neuronal activity using EEG or fMRI(Functional magnetic resonance imaging)( is also emphasized in order to better understand the underlying mechanisms of action. Electrophysiological techniques, such as quantitative electroencephalography (qEEG), provide important information about brain functioning at rest and during sensory stimulation. A large amount of data has demonstrated the presence of some excitability changes in the occipital cortex during the interictal period of migraine patients.While some studies have demonstrated hyperexcitability, only a few studies have been able to document a decrease in occipital excitability. This increase in occipital excitability has recently been recognized as an inhibition phenomenon, and a new term "hyperresponsiveness" in migraine has come into use in the last decade. This hyperexcitability has been demonstrated in many neurophysiological and neuroimaging studies as loss of habituation to recurrent stimuli. Clearly, spectral analysis of different frequency bands of qEEG helps us understand the intrinsic activity of the migraineur brain. Differences in peak latency, amplitude, and synchronization of EEG frequency bands in response to sensory stimulation have been reported in migraine patients compared with healthy subjects. In this study, it is planned to make comparative evaluations in the following months with EEG recordings to be taken before and after simultaneous motor cortex and visual cortex stimulation. In this way, the relationship between anodal and cathodal transcranial direct current stimulation and different frequency bands in the occipital region will be determined by comparing the active treatment and sham groups.

Review studies and recent studies from our country have shown that tDCS treatment is an effective and safe prophylactic treatment in migraine patients with allodynia in both short and long-term follow-ups. In order to obtain better clinical evidence in this field, as emphasized in the Cochrane analysis conducted in 2018; Randomized controlled studies with larger samples and clinically meaningful long-term results are needed. In these studies, it is planned to test the clinical effect of a protocol combination, which has been shown to be particularly effective, in prophylaxis in migraine patients in a large sample group, while also evaluating its neurophysiological responses in active and sham groups.

ELIGIBILITY:
Inclusion Criteria:

* Episodic migraine without aura and with aura, with frequent attacks (>4 or more), diagnosed according to the International Classification of Headache Disorders; The diagnosis must meet the 2018 ICHD-3 criteria for migraine without aura and migraine with aura.
* Patients whose previous prophylactic treatments have failed and who cannot or do not want to use treatments for various reasons
* The duration of the disease must be at least 12 months.
* Not having received any botulinum toxin treatment in the last 3 months
* Having the mental functionality and education to understand the scales used
* Patients who volunteered to participate in the research.

Exclusion Criteria:

* Pregnancy or breastfeeding
* People with clinical evidence of brain damage
* Metallic implant head
* Heart battery
* History of seizures and chronic pain associated with other pathologies
* Other major neurological or major neuropsychiatric diseases;
* Other chronic pain syndromes;
* Other types of primary or secondary headaches;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in headache diary variables | Baseline (Before Treatment) / 1 month and 3 months after treatment
  The number of migraine attacks, pain intensity, duration of each attack and the number of painkillers taken will be evaluated. Patients will answer this diary throughout the entire experimental period (months).

SECONDARY OUTCOMES:
EEG Power Spectrum Analysis | Baseline (Before Treatment) / 1 month and 3 months after treatment
  10 minutes of resting-state EEG recording.EEG data will be separated into one-second epochs after they are cleared of noise. Power spectrums of these data will be obtained in the delta, theta, alpha, beta and gamma frequency bands. Each epoch will be analyzed by Fast Fourier Transform (FFT, Fast Fourier Transform) with 10% Hanning window, then power spectrum analysis will be performed, giving the frequency values for each electrode by averaging all FFTs. Maximum peaks will be determined in the delta (0.5-3.5 Hz), theta (4-7 Hz), alpha (8-13 Hz), beta (15-28 Hz) and gamma (28-48 Hz) frequency bands. these values will be used in statistical analysis for each person and electrode.
EEG Coherence Analysis | Baseline (Before Treatment) / 1 month and 3 months after treatment
  Coherence measurements at delta, theta, alpha, beta and gamma frequencies can be analyzed for either intra-hemispheric electrode connections or inter-hemispheric electrode connections.Coherence values take values between 0-1. Values close to 0 indicate that there is no connection at the determined frequency between the two calculated electrode regions, while values close to 1 indicate a high coupling between the two electrode regions.Coherence values will be calculated with the Brain Vision Analyzer program using the formula below.The data obtained during memory and visualization will be separated into one-second epochs after they are cleared of noise.Power spectrums of these data will be obtained in the delta, theta, alpha, beta and gamma frequency bands. Each epoch will be analyzed by Fast Fourier Transform with 10% Hanning window.Then, these data will be calculated for all possible electrode pairs using the brain vision analysis program with the formula given below.
EEG functional connectivity analysis | Baseline (Before Treatment) / 1 month and 3 months after treatment
  10 minutes of resting-state EEG recording. eLORETA software will be used for functional connectivity analysis. sLORETA /eLORETA is an online free software developed by Roberto Pascual-Marqui and his team (http://www.uzh.ch/keyinst/loreta.htm). eLORETA is an algorithm developed to solve the inverse problem and it does not contain localization bias even in the presence of noise . In this software, resting state data with eyes closed, separated into 2 second epochs, whose artifacts are cleaned by preprocessing, will be used. The relevant areas to be analyzed in the cortical plane and the relevant frequency band gaps will be determined. The time series containing the eLORETA current source density obtained from these areas will be calculated and a "lagged linear coherence" matrix will be created to be applied in graph theory (Vecchio et al., 2014). "Lagged linear coherence" will give correct physiological connectivity unaffected by volume conduction and low spatial resolution.
Changes in the Headache Impact Scale (HIT-6) | Baseline (Before Treatment) / 1 month and 3 months after treatment
  Headache Impact Scale items evaluate vitality, pain, and psychological distress, as well as domains such as sociability, role, and cognitive functioning. Headache Impact Test (HIT-6) questionnaire was designed to helping describe and communicate the way people feel and what they cannot do because of headaches. Interpreting Headache Impact Test scores is achieve through a simple summary of the six items in the survey, ranging from 36 to 78 with larger scores reflecting greater impact. Levels of headache impact severity can be categorized using score ranges based on the HIT-6 interpretation guide into one of four areas: little or no impact (49 or less), some impact (50-55), substantial impact (56-59), and severe impact (60-78).
Changes in Visual Analogue Scale (VAS) | Baseline (Before Treatment) / 1 month and 3 months after treatment
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
  Ask the patient to rate their current level of pain by placing a mark on the line. Use a ruler to measure the distance in centimetres from the 'no pain marker' (or zero) to the current pain mark. This provides a pain intensity score out of 10; for example, 6 out of 10 (or 6/10).
MoCA Tests Scores | Baseline (Before Treatment) / 1 month and 3 months after treatment
  The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Time to administer the MoCA is approximately 10 minutes. The total possible score is 30 points; a score of 26 or above is considered normal.
Beck depression Tests Scores | Baseline (Before Treatment) / 1 month and 3 months after treatment
  The Beck Depression Inventory (BDI; Beck & Steer, 1993) is a 21-item self-report instrument that generates one score reflecting the level of depression as being minimal, mild, moderate, or severe.
Anxiety scales | Baseline (Before Treatment) / 1 month and 3 months after treatment
  Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
tDCS side effect registration form | Baseline (Before Treatment) / 1 month and 3 months after treatment
  Any side effects occurring in the application area (during or after) Any general side effects that occur at the end of the application will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Lütfü Hanoğlu, Prof. DR. MD, Principal Investigator — Medipol University
Locations (1):
- İstanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No